CLINICAL TRIAL: NCT05398718
Title: Bi-directional Real-world Cohort Study on Sotrovimab and Its Impact on the Strength and Duration of the Immune Response to Natural SARS-CoV-2 Infection in Real-life Setting in the UAE and the Kingdom of Bahrain
Brief Title: Study on Sotrovimab and Its Impact on the Immune Response to COVID-19 Infection in Real-life in the UAE and Bahrain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Abu Dhabi Health Services Company (Other Government)
Responsible Party: Sponsor
Other Study IDs: Abu Dhabi Health Services
Record Dates: First submitted 2022-04-29; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: Sotrovimab
MeSH Terms: conditions — COVID-19 | interventions — sotrovimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sotrovimab Arm
  Interventions: Drug: Sotrovimab
- Control

INTERVENTIONS:
Drug: Sotrovimab — collect local clinical evidence for sotrovimab effect in the real-life setting
  Groups: Sotrovimab Arm

SUMMARY:
The United Arab Emirates (UAE), the Kingdom of Bahrain, Kuwait, Oman, and Qatar have authorised sotrovimab for emergency use. Local experience among physicians include recent successful COVID-19 vaccine pivotal studies supported by the authorities' willingness to expedite understanding of the role of monoclonal antibodies such as sotrovimab in the management of COVID-19 and expertise to integrate the latest knowledge into the local or regional COVID-19 management guidelines. The aim of this study is to collect local clinical evidence for sotrovimab effect in the real-life setting in the UAE and the Kingdom of Bahrain. Overall study population is 20,000 and the duration of the study will be approximately six months from recruitment date.

ELIGIBILITY:
Inclusion Criteria:

* Adults and paediatric patients (≥ 12 years of age weighing at least 40 kg)
* Mild-to-moderate COVID-19
* Positive results of direct SARS-CoV-2 viral testing
* High risk for progression to severe COVID-19

Exclusion Criteria:

* Patients who are hospitalised due to COVID-19 before sotrovimab administration
* Patients who require oxygen therapy due to COVID-19 before sotrovimab administration oPatients who received pharmacological treatment including monoclonal antibodies to any components of SARS-CoV-2 virus within 6 months prior to enrolment into the study in retrospective and prospective arms.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with mild-to-moderate COVID-19 as confirmed by approved local laboratory tests
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
• Proportion of patients with COVID-19 progression through Day 29 after sotrovimab administration: | 6 months
  * Proportion of patients with COVID-19 progression through Day 29 after sotrovimab administration:
    * Requiring supplemental oxygen
    * Requiring ICU and/or general ward admission
    * Death
  * Time to first PCR negative status after the COVID-19 symptom onset
  * Time to first PCR negative status after date of sotrovimab administration
To assess the impact of sotrovimab on the strength and duration of the immune response to natural SARS-CoV-2 infection in real-life setting in the UAE and Bahrain. | 6 months
  Defined as
  • Change from baseline in mean levels of elevated SARS-CoV-2 functional neutralising antibodies at Day 29, Day 60 and Day 180 after sotrovimab administration, these will be presented as proportion of patients with that response

SECONDARY OUTCOMES:
To evaluate the impact of sotrovimab on the duration and the severity of COVID-19 clinical symptoms | 6 months
  Time to key clinical symptoms alleviation from symptom onset and sotrovimab administration at baseline, Day 29 after sotrovimab administration and Day of symptoms free (for all 350 patients in the interventional phase and part of the patients in the observational phase). Key clinical symptoms alleviation is defined as the clinical resolution of shortness of breath, fever, and body ache
To evaluate the impact of sotrovimab in reducing SARS-CoV-2 viral load and in preventing COVID-19 respiratory disease progression. | 6 months
To assess the safety of sotrovimab in real-life setting in the UAE and Bahrain | 6 months
  Defined as:
  * Occurrence of adverse events (AEs) and serious adverse events (SAEs) through Day 29 after sotrovimab administration
  * . Proportion of patients with AEs and SAEs through Day 29 after sotrovimab administration.
To assess the impact of sotrovimab on the strength and duration of the immune response to natural SARS-CoV-2 infection in real-life setting in the UAE and Bahrain. | 6 months
  Defined as:
  • Change from baseline in mean levels of elevated SARS-CoV-2 functional neutralising antibodies at Day 29, Day 60 and Day 180 after sotrovimab administration in patients, who received their complete or incomplete vaccination course within 3 months prior to COVID-19 symptom onset, these will be presented as proportion of patients with that response.

OTHER OUTCOMES:
To evaluate the impact of sotrovimab on incidence and duration of time for supplemental oxygen, length of stay (LOS) in the intensive care unit (ICU), and total hospital LOS. | 6 months
  Defined as:
  Proportion of COVID-19 patients who had ER visits for management of illness, for requirement of supplemental oxygen and/or ICU admission through Day 29 after sotrovimab administration.
Quality of life of patients infused with Sotrovimab | 6 months
  Defined as Change from baseline in health-related quality of life at Day 29 after sotrovimab administration according to the 20-item short form (SF-20) questionnaire (where available / in a selected fraction of patients only in the prospective arm).
  The questionnaire contains items on physical functioning, role functioning, social functioning, mental health, health perception and pain, the score of all measures is transformed linearly to 0-100 scales, with 0 and 100 assigned to the lowest and highest possible scores, respectively. a high score indicates better health
To evaluate the clinical impact of sotrovimab in preventing mortality. | 6 months
  Defined as All-cause mortality during 29 days after sotrovimab administration

CONTACTS AND LOCATIONS:
Locations (1):
- The National Taskforce for combating COVID-19, Royal Medical Services., Manama, Bahrain

IPD SHARING:
Plan to Share IPD: No